CLINICAL TRIAL: NCT03552380
Title: A Phase II Study to Evaluate the Safety, Pharmacodynamics, and Efficacy of Entinostat in Combination With Nivolumab Plus Ipilimumab in Patients With Renal Cell Carcinoma Previously Treated With Nivolumab Plus Ipilimumab
Brief Title: Study of Entinostat With Nivolumab Plus Ipilimumab in Previously Treated Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder halted development of compound in this disease
Sponsor: Roberto Pili (Other)
Collaborators: Bristol-Myers Squibb (Industry); Syndax Pharmaceuticals (Industry); Indiana University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Roberto Pili, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU17-326
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — entinostat; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entinostat, Nivolumab and Ipilimumab (Experimental): Entinostat: 5mg, 3mg, or 2mg orally (PO) on D1, 8, 15 plus Nivolumab: 3 mg/kg IV D1 and Ipilimumab 1 mg/kg IV D1
  Each cycle is 21 days
  Interventions: Drug: Entinostat; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Entinostat — RP2D will be determined with a 6 patient safety lead-in. Entinostat will continue until disease progression or prohibitive toxicity. Cycles 1-4 are 21 day cycles. Cycles 5 and subsequent are 28 day cycles.
  Other Names: MS-275; SND-275
Drug: Nivolumab — Nivolumab will continue until disease progression or prohibitive toxicity. Cycles 1-4 are 21 day cycles. Cycles 5 and subsequent are 28 day cycles.
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab will be administered in combination with entinostat and nivolumab for Cycles 1-4 only.
  Other Names: Yervoy

SUMMARY:
This is a Phase II, open-label, safety, pharmacodynamic and efficacy study of entinostat in combination with nivolumab and ipilimumab in subjects with metastatic renal cell carcinoma (RCC) who have progressed on ipilimumab + nivolumab regimen. Prior to Phase II, a safety lead-in will be conducted to establish the RP2D of entinostat when used in combination with ipilimumab + nivolumab. Subjects will initially be treated with the combination of oral entinostat and intravenous (IV) nivolumab plus ipilimumab. Entinostat will be dosed weekly, and nivolumab and ipilimumab will be dosed every 3 weeks, for a total of four, 3-week cycles. Following these first four cycles, entinostat will continue to be administered weekly in combination with nivolumab every 4 weeks or every 2 weeks based on subject tolerance (ipilimumab will be discontinued), with treatment continued until disease progression or prohibitive toxicity. Anti-tumor activity will be assessed by radiological tumor assessments conducted at baseline and every 6 weeks thereafter using RECIST version 1.1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 within 28 days prior to registration.
* Histological or cytological evidence of renal cell carcinoma (initial diagnosis).
* Metastatic disease
* Progressive disease (PD) on nivolumab + ipilimumab regimen. Note: Patients who have completed at least one dose of ipilimumab + nivolumab and progress or have completed the 4 doses of ipilimumab + nivolumab and progress during nivolumab monotherapy maintenance are eligible unless they have received additional treatment(s) for their renal cell carcinoma prior to registration. Patients who discontinue prior ipilimumab + nivolumab or nivolumab monotherapy for toxicity are excluded. Patients who receive nivolumab or other anti-PD-1/PD-L1 agents as subsequent therapy after ipilimumab + nivolumab are excluded.
* Target lesions according to RECIST v1.1 or non-target bone lesions assessed by bone scan or positron emission tomography (PET) scan.
* A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration, have been off corticosteroids for ≥ 4 weeks, and are asymptomatic.
* Prior cancer treatment (excluding nivo/ipi) must be completed at least 28 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia or neuropathy) to ≤Grade 1 or baseline. If subject underwent major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
* Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 28 days prior to registration

  * Platelets ≥100 x 10^9/L
  * Absolute Neutrophil Count (ANC) ≥1.5 x 10^9/L
  * Hemoglobin (Hgb) ≥9 g/dL or ≥5.6 mmol/L
  * Creatinine OR Measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of CrCl) Creatinine clearance should be calculated per institutional standard ≤1.5 x the upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels >1.5 x institutional ULN
  * Bilirubin ≤1.5 x ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
  * Aspartate aminotransferase (AST) ≤3 x ULN
  * Alanine aminotransferase (ALT) ≤3 x ULN
  * International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT/INR/PTT is within therapeutic range of intended use of anticoagulants
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test during screening and a negative urine pregnancy test within 3 days prior to first dose of study drug. If the screening serum test is done within 3 days prior to receiving the first dose of study drug, a urine test is not required.
* Women of childbearing potential must be willing to abstain from heterosexual intercourse or to use an effective method of contraception from the time of informed consent until 5 months after the last dose of study drug.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving study drugs and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 3 months after the last dose of entinostat.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
* Life expectancy of at least 6 months per investigator discretion.

Exclusion Criteria:

* Subjects meeting any of the criteria below may not participate in the study:

  * History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including, but not limited to:

    * Myocardial infarction or arterial thromboembolic events within 6 months prior to screening or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a corrected QT interval (QTc) interval > 470 msec.
    * Uncontrolled hypertension or diabetes mellitus.
    * Another known malignancy that is progressing or requires active treatment.
    * Any prior history of other cancer within the prior 5 years with the exception of adequately treated basal cell carcinoma or cervical intraepithelial neoplasia [CIN]/cervical carcinoma in situ or melanoma in situ).
    * Active infection requiring systemic therapy.
    * Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
  * Pregnant or breastfeeding. Note: breast milk cannot be stored for future use while the mother is being treated on study.
  * Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
  * Allergy to benzamide or inactive components of entinostat.
  * Hypersensitivity to nivolumab, ipilimumab, or any of their excipients.
  * Treatment with any investigational drug or device within 4 weeks prior to registration.
  * Treatment with systemic steroids within 4 weeks prior to registration. Note: adrenal replacement doses of steroids (for example prednisone 10mg daily) are permitted while on study.
  * Evidence of active autoimmune disease requiring systemic treatment within the past 90 days or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
  * Interstitial lung disease or history of pneumonitis requiring treatment with corticosteroids.
  * Diagnosis of immunodeficiency; or is receiving chronic systemic corticosteroid therapy or other immunosuppressive therapy (excludes inhaled corticosteroids) within 4 weeks prior to registration.
  * Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies). Testing during screening is not required.
  * Known active hepatitis B (e.g., hepatitis B surface antigen-reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]). Subjects with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA test must be performed in these subjects prior to study treatment, and results must be negative to be eligible. Subjects with a history of hepatitis C must be tested for presence of hepatitis C virus (HCV) antibody. If HCV antibody positive, subjects will only be eligible if polymerase chain reaction is negative for HCV RNA.
  * Has received a live vaccine within 30 days prior to planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, MD, Principal Investigator — Indiana Univervisty Simon Cancer Center
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Indiana Univeristy Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab: Patients received oral entinostat at a dose of 5 mg every 7 days continuously with nivolumab at a dose of 3 mg/kg mg IV every three weeks in combination with ipilimumab at a dose of 1 mg/kg every 3 weeks X 4 doses. Then, nivolumab 480 mg was continued every 4 weeks.
- Phase II, Dose Level 2 : Entinostat 3 mg With Nivolumab and Ipilimumab: Patients received oral entinostat at a dose of 3 mg every 7 days continuously with nivolumab at a dose of 3 mg/kg mg IV every three weeks in combination with ipilimumab at a dose of 1 mg/kg every 3 weeks X 4 doses. Then, nivolumab 480 mg was continued every 4 weeks.
Period: Study Treatment
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2 : Entinostat 3 mg With Nivolumab and Ipilimumab
Started | 5 | 7
Completed | 0 | 1
Not Completed | 5 | 6
Not completed — Disease Progression | 3 | 4
Not completed — Adverse Event | 2 | 2
Period: Follow up
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2 : Entinostat 3 mg With Nivolumab and Ipilimumab
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 5 | 7
Completed | 0 | 0
Not Completed | 5 | 7
Not completed — PI request to move remaining patients on follow-up to Off study | 2 | 2
Not completed — Death | 3 | 4
Not completed — Site IRB terminated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab: Patients received oral entinostat at a dose of 3 mg every 7 days continuously with nivolumab at a dose of 3 mg/kg mg IV every three weeks in combination with ipilimumab at a dose of 1 mg/kg every 3 weeks X 4 doses. Then, nivolumab 480 mg was continued every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Onology group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Onology group (ECOG) Performance Status is described as follows:
  0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    ECOG = 0 | 3 | 4 | 7
    ECOG = 1 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Via RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From C1D1 until death or up to 31 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase II, Dose Level 1:Entinostat 5 mg With Nivolumab and Ipilimumab: Patients received oral entinostat at a dose of 5 mg every 7 days continuously with nivolumab at a dose of 3 mg/kg mg IV every three weeks in combination with ipilimumab at a dose of 1 mg/kg every 3 weeks X 4 doses. Then, nivolumab 480 mg was continued every 4 weeks.
Arm/Group | Phase II, Dose Level 1:Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab
Number analyzed (Participants) | 5 | 7
percentage of participants | 20 [5.1 to 71.6] | 42.9 [9.9 to 81.6]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Assess adverse events according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4
Time Frame: From C1D1 until death or up to 31 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab
Number analyzed (Participants) | 5 | 7
Participants
  Number of patients had at least one adverse event of any grade. | 5 | 7
  Number of patients had at least one grade 3 or greater adverse event. | 5 | 3
  Number of patients had at least one grade 3 or greater treatment related adverse event | 5 | 2
  Number of patients having serious adverse event. | 3 | 3

3. Secondary Outcome: Objective Response Rate Via Immune Related Response Criteria (irRC)
Description: Per immune-related response criteria (irRC): Complete Response(irCR), Disappearance of all target and nontarget lesions; Partial Reponse (irPR), ≥ 50% decrease in tumor burden compared with baseline; Progressive Disease (irPD), >= 25% increase in tumour burden relative to nadir or the appearance new lesions; Stable Disease (irSD), not meeting criteria for irCR or irPR, in absence of irPD. Overall Response (OR) = irCR + irPR
Time Frame: From C1D1 until death up to 31 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab
Number analyzed (Participants) | 5 | 7
Percentage of participants | 20 [5.1 to 71.6] | 28.6 [3.7 to 71]

4. Secondary Outcome: Progression Free Survival (PFS) Via RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  PFS is defined as time from starting treatment to disease progression met by RECIST 1.1 or death as a result of any cause.
Time Frame: Up to 31 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab
Number analyzed (Participants) | 5 | 7
months | 4.3 [1.3 to NA] — Upper limit was not reached due to an insufficient number of participants with events. | 11.7 [1.9 to NA] — Upper limit was not reached due to an insufficient number of participants with events.

5. Secondary Outcome: Progression Free Survival (PFS) Via irRC
Description: Per immune-related response criteria (irRC): Complete Response(irCR), Disappearance of all target and nontarget lesions; Partial Reponse (irPR), ≥ 50% decrease in tumor burden compared with baseline; Progressive Disease (irPD), >= 25% increase in tumour burden relative to nadir or the appearance new lesions; Stable Disease (irSD), not meeting criteria for irCR or irPR or irPD.
  PFS is defined as time from starting treatment to disease progression met by irRC or death as a result of any cause.
Time Frame: Up to 31 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab
Number analyzed (Participants) | 5 | 7
months | 4.3 [1.3 to NA] — Upper limit was not reached due to an insufficient number of participants with events. | 11.7 [5.9 to NA] — Upper limit was not reached due to an insufficient number of participants with events.

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined from Day 1 of treatment until death as a result of any cause
Time Frame: Up to a maximum of 59 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab
Number analyzed (Participants) | 5 | 7
months | 49.9 [6.7 to NA] — Upper limit was not reached due to an insufficient number of participants with events. | 36 [5.9 to NA] — Upper limit was not reached due to an insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 59 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 31 months.
Description: Adverse events were collected for every subject at every cycle of treatment (14 cycles). First 4 cycles at an interval of 21 days and rest at an interval of 28 days from the time of consent until 100 days after last treatment. Serious adverse events were reported from time of signed informed consent until 100 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first.
Arm/Group | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 3/5 | 4/7
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/7
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab (N=5) | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab (N=7)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II, Dose Level 1: Entinostat 5 mg With Nivolumab and Ipilimumab (N=5) | Phase II, Dose Level 2: Entinostat 3 mg With Nivolumab and Ipilimumab (N=7)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 5 (6)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (5) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (6) | 3 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (4)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT03552380/Prot_SAP_001.pdf